CLINICAL TRIAL: NCT04422145
Title: Hypoglycemia Requiring Emergency Services Intervention: Patient Characteristics, Outcome and Cardiovascular Risk Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Yorkshire Ambulance Service NHS Trust (Other Government); LifeScan (Industry)
Responsible Party: Principal Investigator, Ramzi Ajjan, Professor of metabolic medicine, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P1
Record Dates: First submitted 2020-05-13; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia | interventions — Standard of Care

STUDY DESIGN:
Masking Description: Due to the nature of the intervention 9a nurse led education programme) it was not possible to mask participant or trial team to the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interventional/intensive (Active Comparator): Participants received a structured nurse led education programme surrounding hypoglycaemia. They were encouraged to use self monitoring of blood glucose (SMBG) and had their diabetes medications adjusted according to this. They also received information on how to avoid hypoglycaemia (including the effects of diet, exercise, alcohol and their medications) and how to treat hypoglycaemia should it occur.
  Interventions: Behavioral: Structured nurse led intervention programme
- Standard (Placebo Comparator): Participants returned to their standard diabetes care provider with no intervention.
  Interventions: Other: Standard care
- Observational (No Intervention): Participants were happy to have baseline characteristics collected and be followed up using electronic records in a longitudinal fashion but did not wish to be randomized. The observational and standard groups therefore received the same diabetes care.

INTERVENTIONS:
Behavioral: Structured nurse led intervention programme — A diabetes research nurse, over a period of 12 months, provided a structured education programme to participants focussing on the avoidance of hypoglycaemia and the treatment of this if/when it occurred.
  Arms: Interventional/intensive
Other: Standard care — Participants continue on their current diabetes care plan and are looked after by their usual diabetes care provider
  Arms: Standard

SUMMARY:
Patients who suffer hypoglycaemia in the community requiring the services of an ambulance are known to have a high short term mortality based on previous work. What is not known is the demographics of this group and also what the cause of death was for individuals whom unfortunately passed away in the time following ambulance callout. Importantly, studies looking at interventions to reduce poor outcomes in this group are lacking. The investigators conducted a pilot trial with the main goals to:

1. Characterise this group in more detail and ascertain what was recorded as cause of death in those whom passed away in the months/years following community hypoglycaemia
2. Ascertain if a simple nurse led intervention, focusing on educating participants on avoidance of hypoglycaemia, could improve outcome.

DETAILED DESCRIPTION:
Previous studies, including our own, have shown that in those with diabetes, severe hypoglycaemia (defined as requiring the assistance of emergency ambulance in the community) carries with it a high mortality in the immediate months/short years following the event. What isn't known is what this group of patients dies of and what the demographics of this group may be. This is important as this is a vulnerable patient group in whom few interventions to reduce this excess mortality have been trialled.

Through a collaboration with a local ambulance service, the hospital diabetes research team set out to recruit participants to a small, pilot, randomized controlled trial to try and ascertain more about the demographics of this group, follow them up in a longitudinal fashion and report on their causes of death using information recorded on death certificates (a statutory requirement in the UK). Additionally the investigators sought to provide pilot data on whether a structured nurse led intervention programme could reduce risk.

The local ambulance service contacted the research team, with patient consent, once they had been called to treat a patient with diabetes whom had severe hypoglycaemia. Within 7 days a research nurse approached those whom had given consent to invite them to take part in a clinical trial. Full eligibility criteria are available elsewhere in this document. Following this, groups were split in the following way:

1. Intensive group - participants were randomized to receive a structured nurse led intervention aiming to educate them on the treatment of and how to avoid hypoglycaemia.
2. Standard group - participants were randomized to continue on their current diabetes treatment and were returned to their standard diabetes care provider.
3. Observational group - participants were happy to have a baseline visit, and for their case to reviewed using electronic records moving forward, but they did not wish to be randomized to an intervention.

All three groups had baseline data collected including:

* Diabetes specific information, including HbA1c, type of diabetes, diabetes therapy, duration of diabetes, presence of complications. Blood tests were taken at baseline for all groups if participants consented to have this done.
* Demographic data - including age, gender, smoking status, BMI
* Information of co-morbidity - Any other illness the participant may suffer from, any medications they take.

Information regarding baseline characteristics was confirmed using electronic patient records.

Those whom were randomized to a nurse led intervention received a structured education programme for 12 months, with the bulk of the work coming in the first 12 weeks.

At 12 months, all participants active engagement in the programme was terminated. Data was collected electronically on new hospital admissions and deaths over this period as well as changes in HbA1c. Participants also had their electronic records screened at study termination and thus data could be provided on outcome at 12 months and study end (in this case 42.6 months.)

ELIGIBILITY:
Inclusion Criteria:

Diabetes mellitus Can provide written informed consent

Exclusion Criteria:

Hypoglycaemia from cause not related to diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
All cause mortality at study endpoint with each participant having a minimum follow up of 12 months and the final analysis of data being done 58 months after the first participant was recruited (this is study endpoint.) | Through study endpoint, which was 58 months following the recruitment of the first participant and 12 months following the recruitment of the last participant.
  Electronic review of participants records to ascertain if they had passed away during the study

SECONDARY OUTCOMES:
All cause mortality at 12 months from recruitment. | 12 months
  Assessment of all-cause mortality at 12 months from recruitment to study.
Analyse cause of death at study endpoint (12 months following recruitment of last participant). | Study end point defined as 12 months following recruitment of last participant (approximately 40 months from start of study).
  Using death certificates to compare cause of death between study groups and between type 1 and type 2 diabetes. After cause of death was obtained, participants were grouped into categories as to mortality, eg cardiovascular cause.
Assessment of differences in mortality rate between type 1 and type 2 diabetes participants | Study endpoint (12 months following recruitment of last participant.)
  To analyse mortality at studies endpoint (defined as 12 months following recruitment of last participant)

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Ajjan, PHD, Principal Investigator — Professor of metabolic medicine
Locations (1):
- Diabetes centre, St James hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to do so is currently in place. Of course once data is submitted if other researchers contact us we would consider providing data for the purpose of meta analysis

REFERENCES:
- [Derived] Pearson SM, Whittam B, Kulavarasalingam K, Mitchell-Gears A, James C, Ajjan RA. Reduction in cardiovascular mortality following severe hypoglycemia in individuals with type 2 diabetes: the role of a pragmatic and structured intervention : Structured intervention for community hypoglycemia. Cardiovasc Diabetol. 2021 Jan 12;20(1):18. doi: 10.1186/s12933-020-01204-3. PMID 33435992

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04422145/Prot_SAP_000.pdf